CLINICAL TRIAL: NCT02124564
Title: Multicenter, Open-Label, Long-Term Study to Investigate the Safety of Conversion to Lacosamide at Doses up to 600 mg/Day as Monotherapy in Japanese Adults With Partial-Onset Seizures With or Without Secondary Generalization
Brief Title: A Trial to Evaluate the Long Term Safety and Tolerability of Lacosamide Taken as Monotherapy in Adults With Partial-onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0057
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Epilepsy; Partial-onset Seizures
Keywords: Lacosamide; Epilepsy; Focal, Partial-Onset Seizures with or without secondary generalization; Monotherapy
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): Open-label, single-arm
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Lacosamide (LCM) immediate-release, film-coated tablets at a strength of 50 mg orally administered twice daily in two equally divided doses.
  * 4-week Titration Period: Starting on LCM 100 mg/day increased by 100 mg/day each week until 400 mg/day dose reached at the beginning of Week 4 .
  * The AED Withdrawal Period and Monotherapy Period (52- week Evaluation Period plus a Follow Up Period): During the AED Withdrawal and Monotherapy Period, the investigator may increase or decrease the dose of LCM to optimize tolerability and seizure control. The LCM dose may be decreased no lower than 200 mg/day or increased, no faster than 100 mg/day per week, up to 600 mg/day.
  Other Names: Vimpat

SUMMARY:
This study is to evaluate the long-term safety and tolerability of Lacosamide (LCM) 200 mg/day to LCM 600 mg/day taken in monotherapy in Japanese subjects who currently have partial-onset seizures with or without secondary generalization and who are treated with a single Anti-Epileptic Drug (AED) with marketing approval in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and ≥16 years of age
* Subject has a diagnosis of epilepsy, having experienced unprovoked partial-onset seizures (IA, IB, or IC with clear focal origin) that are classifiable according to the International League Against Epilepsy (ILAE) Classification of Epileptic Seizures, 1981
* Subject experiences partial-onset seizures despite appropriately chosen and adequately tried treatment with 1 antiepileptic drug (AED)
* Subject has been treated for epilepsy with a stable dose of 1 marketed AED The use of benzodiazepines is permitted as rescue therapy for epilepsy. Benzodiazepines may have been used as needed but not more frequently than once per week.

Exclusion Criteria:

* Subject has a history or presence of seizures of other types than partial onset (IA, IB, or IC with clear focal origin)
* Subject is taking benzodiazepines for a nonepilepsy indication (Exception: Concomitant use of benzodiazepines is allowed if the subject is taking them on a regular basis, has been on a stable dose for at least 1 month prior to Visit 1, and does not require changes in the dosage and administration throughout the study period. However, concomitant use of benzodiazepines on an as needed basis is not permitted.)
* Female subject who is pregnant or nursing, and/or a woman of childbearing potential who is not surgically sterile, 2 years postmenopausal or does not practice 1 highly effective method of contraception, unless sexually abstinent, for the duration of the study
* Female subject of childbearing potential taking enzyme-inducing antiepileptic drugs (EI-AEDs: CBZ, phenytoin, barbiturates, primidone, topiramate) who is not surgically sterile, 2 years postmenopausal or does not practice 1 highly effective method of contraception according to the World Health Organization (WHO) recommendation (ie, depot medroxyprogesterone acetate, norethisterone enantate, intrauterine devices, combined injectables, and progestogen implants) with administration of EI-AEDs or does not practice 2 combined methods of contraception (ie, combined hormonal contraception plus barrier method with spermicidal agent), unless sexually abstinent, for the duration of the study
* Subject has sick sinus syndrome without a pacemaker, or a second or third degree atrioventricular (AV) block, or subject has any other clinically relevant electrocardiogram (ECG) abnormalities
* Subject has a history of convulsive status epilepticus within the last 12 months prior to Visit 1

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (11):
- Japan (11):
  - 5, Asaka
  - 1, Hamamatsu
  - 11, Itami
  - 6, Kagoshima
  - 7, Kamakura
  - 10, Nagoya
  - 12, Saitama
  - 8, Sapporo
  - 13, Shinagawa City
  - 4, Shizuoka
  - 9, Toyonaka

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in April 2014 and concluded in November 2017.
Pre-assignment Details: Participant flow refers to Safety Set including all subjects which took at least one dose of study medication.
Groups:
- Lacosamide: Subjects randomized in this arm received lacosamide from 200 mg/day to 600 mg/day, from the Titration to the End of Study Visit (up to 3.5 years).
Period: Treatment Period
Arm/Group | Lacosamide
Started | 19
Started Treatment Period | 19
Started Titration Period | 19
Started AED Withdrawal Period | 19
Started Monotherapy Period | 17
Started Evaluation Period | 17
Started Follow-Up Period | 13
Completed | 12
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 2
Period: Taper Period
Arm/Group | Lacosamide
Started (Subjects receiving LCM >200mg/day at the End-of-Study/Early Withdrawal Visit should be tapered off.) | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refer to the Safety Analysis Set which included all subjects who took at least 1 dose of study drug.
Arm/Group | Lacosamide
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Japanese) | 19
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Incidence of Treatment-Emergent Adverse Events (TEAEs) During the Study
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From the Titration Period (investigational product is taken) to the End of Study Visit (up to 3.5 years)
Measure: Count of Participants; unit: Participants
Groups:
- Lacosamide (Safety Set): Subjects randomized in this arm received lacosamide from 200 mg/day to 600 g/day, from the Titration to the End of Study Visit (up to 3.5 years).
Arm/Group | Lacosamide (Safety Set)
Number analyzed (Participants) | 19
Participants | 19

2. Primary Outcome: Number of Subjects Who Withdraw Due to Adverse Events (AEs) During the Study
Description: as for outcome 1
Time Frame: From the Titration Period (investigational product is taken) to the End of Study Visit (up to 3.5 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide (Safety Set)
Number analyzed (Participants) | 19
Participants | 2

3. Primary Outcome: Number of Subjects With at Least One Incidence of Serious Adverse Events (SAEs) During the Study
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is as infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above
Time Frame: From the Titration Period (investigational product is taken) to the End of Study Visit (up to 3.5 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide (Safety Set)
Number analyzed (Participants) | 19
Participants | 2

4. Secondary Outcome: Number of Subjects Remaining Seizure Free for 6 Consecutive Months During the Monotherapy Period
Description: Subjects were considered seizure free if their seizure counts for every day over the entire Treatment Period was zero and if they completed the Treatment Period.
  A subject was considered seizure free, if no seizure occurred during the 6 consecutive months in the Evaluation Period. If one of the following occurred, the subject was not considered seizure free:
  * A documented seizure during 6 consecutive months of the Evaluation Analysis Period
  * Subject discontinued the study prematurely during the Evaluation Analysis Period
  * Missing Seizure Count Case Report Forms (CRFs) prior to completing the Evaluation Analysis Period
Time Frame: From the beginning of the Monotherapy Period to the end of the Follow-Up Period (up to 3.1 years until the time of approval granted)
Population: The Full Analysis Set (FAS) consisted of subjects in the Safety Set (SS) who had at least 1 seizure diary assessment. Subjects who discontinued before the end date of 6 consecutive months were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Lacosamide (FAS): Subjects randomized in this arm received lacosamide from 200 mg/day to 600 mg/day, from the Titration to the End of Study Visit (up to 3.5 years).
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 13
Participants | 6

5. Secondary Outcome: Number of Subjects Remaining Seizure Free for 12 Consecutive Months During the Monotherapy Period
Description: Subjects were considered seizure free if their seizure counts for every day over the entire Treatment Period was zero and if they completed the Treatment Period.
  A subject was considered seizure free, if no seizure occurred during the 12 consecutive months in the Evaluation Period. If one of the following occurred, the subject was not considered seizure free:
  * A documented seizure during 6 consecutive months of the Evaluation Analysis Period
  * Subject discontinued the study prematurely during the Evaluation Analysis Period
  * Missing Seizure Count Case Report Forms (CRFs) prior to completing the Evaluation Analysis Period.
  Subjects who discontinued before the end date of 6 consecutive months were included in this analysis.
Time Frame: as for outcome 4
Population: The Full Analysis Set (FAS) consisted of subjects in the SS who had at least 1 seizure diary assessment. Subjects who discontinued before the end date of 12 consecutive months were included in this Analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 13
Participants | 6

6. Secondary Outcome: Percentage of Participants in the Monotherapy Period Without Discontinuation Due to Adverse Events (AE) or Lack of Efficacy (LOE)
Description: For Time to discontinuation (event), Retention rate and 95% CI was calculated using the Kaplan-Meier method. Retention rate is indicated in Percent and 95% confidence intervals (CI) with respect to the Time to discontinuation.
Time Frame: as for outcome 4
Population: The Full Analysis Set (FAS) consisted of subjects in the Safety Set (SS) who had at least 1 seizure diary assessment. Subjects who discontinued before Monotherapy Period were not included in this Analysis.
Measure: Median (95% Confidence Interval); unit: Percentage of participant
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 17
Percentage of participant
  Retention Rate after 6-months | 81.3 [52.46 to 93.54]
  Retention Rate after 12-months | 81.3 [52.46 to 93.54]
  Retention Rate after 18-months | 81.3 [52.46 to 93.54]
  Retention Rate after 24-months | 81.3 [52.46 to 93.54]

7. Secondary Outcome: Plasma Concentrations of Lacosamide Versus Time Postdose
Description: Dose-normalized lacosamide Plasma Concentration (µg/mL) by Visit and Dose during the Evaluation Period.
Time Frame: From Titration Period up to Week 94
Population: Two Subjects withdrew during the AED Withdrawal Period (prior to the Evaluation Period).
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Lacosamide (Safety Set)
Number analyzed (Participants) | 17
µg/mL
  Concentration at First Visit | 0.028 (0.016)
  Concentration at Last Visit | 0.034 (0.010)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Visit 1 until Safety Follow-Up Visit (up to week 2 after last dose), for approximately 3.5 years
Arm/Group | Lacosamide
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=19)
Convulsion (Nervous system disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Lacosamide (N=19)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (5)
Dry eye (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (13)
Influenza (Infections and infestations) | 2 (2)
Acute tonsillitis (Infections and infestations) | 1 (2)
Bronchitis (Infections and infestations) | 1/16 (1)
Cystitis (Infections and infestations) | 1 (2)
Herpes virus infection (Infections and infestations) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (4)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Heat illness (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood growth hormone increased (Investigations) | 1 (1)
Crystal urine present (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (2)
White blood cell count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pubic pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 10 (13)
Somnolence (Nervous system disorders) | 8 (9)
Headache (Nervous system disorders) | 3 (5)
Tremor (Nervous system disorders) | 2 (2)
Cerebellar ataxia (Nervous system disorders) | 1 (1)
Complex partial seizures (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Simple partial seizures (Nervous system disorders) | 1 (1)
Sudden onset of sleep (Nervous system disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3)
Chloasma (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2013-10-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT02124564/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT02124564/SAP_001.pdf